CLINICAL TRIAL: NCT02900638
Title: Pilot Study of Physical Health Effects of Cities Mentor Project
Brief Title: Health Effects of Mentoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Edith Chen, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00203223
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Health
Keywords: mentoring; children; cardiovascular health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Mentor/Mentee) (Experimental)
  Interventions: Behavioral: Mentoring
- Wait list control (No Intervention)

INTERVENTIONS:
Behavioral: Mentoring — Youth in the intervention group will participate in one-on-one mentoring sessions (between mentors and mentees) once per week after school. Mentoring sessions will focus on the development of a social bond between mentor and mentee.
  Arms: Intervention (Mentor/Mentee)

SUMMARY:
The purpose of this study is to determine whether mentoring is associated with beneficial cardiovascular health effects in both mentors and mentees.

DETAILED DESCRIPTION:
Participants are randomly assigned to either being a mentor or a wait list control. These participants are drawn from a population of undergraduate students. Participants are also randomly assigned to either being a mentee or a wait list control. These participants are drawn from a population of Chicago Public School children. In total, there will be 30 mentors, 30 control mentors, 30 mentees, and 30 control mentees. Participants will come for a laboratory visit in which cardiovascular health measures will be taken (details below). Visits will occur once at baseline (before the intervention starts), and once post-intervention. The protocol will be the same at the two study visits. Participants in the intervention group will engage in one-on-one mentoring sessions (between mentors and mentees) once a week after school for the school year

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student for mentors.
* Chicago Public School student for mentees.

Exclusion Criteria:

* Younger than 9 or older than 14 for mentee conditions.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Obesity [body mass index] | Change in body mass index from baseline to 8 months
  BMI in kg/m^2, weight in kilograms, height in meters
Blood Pressure | Change in blood pressure from baseline to 8 months
Pro-inflammatory cytokines [standardized and averaged value of pro-inflammatory cytokines and CRP] | Change in cytokine composite score from baseline to 8 months
Cholesterol | Change in cholesterol from baseline to 8 months
HbA1c | Change in HbA1c from baseline to 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States